CLINICAL TRIAL: NCT05390697
Title: Educational Videos to Address Vaccine Hesitancy in Childhood Immunization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Prof. Hartono Gunardi, MD, PhD, Professor, Indonesia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1042/UN2.F1/ETIK/PPM.00.02
Record Dates: First submitted 2022-05-16; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Vaccination Refusal; Vaccine Hesitancy
Keywords: health education; health promotion; Indonesia; vaccination; vaccination hesitancy
MeSH Terms: conditions — Vaccination Refusal; Vaccination Hesitancy; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The educational videos included five modules distributed over five weeks.
  Interventions: Other: Educational videos
- Control group (No Intervention): Participants in the control group were given exposure to the digital version of the MCH handbook, 2020 edition, consisting of animated pictures and simple instructions.

INTERVENTIONS:
Other: Educational videos — Educational videos include (1) danger and prevention of VPD; (2) rationales of completing immunization; (3) immunization amid the COVID-19 pandemic; (4) vaccine misconception; and (5) adverse events following immunization and how to treat it. Each video was less than 2 minutes with clear and straightforward messages according to the National Institute of Health guideline for health education. Materials were distributed through WhatsApp and viewed for five weeks.
  Arms: Intervention group

SUMMARY:
Vaccine hesitancy and the COVID-19 pandemic may threaten immunization coverage in children. This study aimed to evaluate the tailored educational videos to reduce vaccine hesitancy and analyze immunization completeness status. The investigators conducted an interventional quasi-experimental study in three subdistricts of North Jakarta, Indonesia. Participants were allocated into the intervention and control groups, and the Parent Attitudes about Childhood Vaccines (PACV) questionnaire was used to assess vaccine hesitancy status before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Parents with children aged 10-18 months
* Parents who had electronic devices that could play videos, such as smartphones or tablets
* Registered in the community health centers database.

Exclusion Criteria:

* Children had contraindicated for immunization
* Children were dropped out if they did not finish their studies.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
The Parent Attitudes about Childhood Vaccines (PACV) Questionnaire | Five weeks after intervention
  Improvement in vaccine hesitancy among Indonesian parents who underwent educational videos intervention, compared to the maternal and child health (MCH) handbook digital version as a standard educational tool

SECONDARY OUTCOMES:
Childhood routine immunization status | Five weeks after intervention
  Childhood routine immunization status (complete/incomplete/improved)

CONTACTS AND LOCATIONS:
Overall Officials: Hartono Gunardi, MD, PhD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Dr. Cipto Mangunkusumo Hospital, Jakarta Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided